CLINICAL TRIAL: NCT04042259
Title: Delayed Primary Closure Using Negative Pressure Wound Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Colleen M Trevino PhD, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00032783
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Infection Abdominal
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Negative Pressure Wound Therapy (Active Comparator): Standardized wound closure with negative pressure therapy.
  Interventions: Device: Abthera
- Historic Cohort (Other): Historic cohort have undergone a midline laparotomy and managed with an open abdomen for at least one day and have contaminated or dirty wound classification.
  Interventions: Procedure: Open adbdomen for post-laparotomy without NPWT device

INTERVENTIONS:
Device: Abthera — Negative Pressure Wound Therapy Device
  Other Names: VERAFLO; Prevena
  Arms: Negative Pressure Wound Therapy
Procedure: Open adbdomen for post-laparotomy without NPWT device — Historic cohort treatment of open abdomen for dirty wounds without use of negative pressure therapy device
  Arms: Historic Cohort

SUMMARY:
Surgical site infection rates for contaminated or dirty laparotomy wounds can be as high as 45%. Surgical management of dirty and contaminated wounds has been controversial in the literature and between surgeons. Primary closure (PC) of these wounds can lead to multiple complications including surgical site infection (SSI), necrotizing soft tissue infection, wound and fascial dehiscence, evisceration, sepsis and hernia development. However, an alternative technique of utilizing secondary intention results in prolonged healing time and increased cost and healthcare resource utilization. Delayed primary closure (DPC) was developed to address many of these issues. Bhangu completed a systematic review and meta-analysis comparing primary versus delayed primary skin closure in contaminated and dirty abdominal wounds. They included 8 studies randomizing 623 patients with contaminated or dirty abdominal wounds to either DPC or PC. The most common diagnosis was appendicitis (77.4%), followed by perforated abdominal viscus (11.5%), ileostomy closure (6.5%), trauma (2.7%), and intra-abdominal abscess/other peritonitis (1.9%). The time to first assessment for DPC was between 2 and 5 days postoperatively. In all studies, the DPC group had significantly less SSIs using a fixed-effect model (odds ratio, 0.65; 95%CI, 0.40-0.93; P = .02). However, heterogeneity was high (72%), and using a random-effects model, the effect was no longer significant (odds ratio, 0.65; 95% CI, 0.25-1.64; P = .36). Additionally, all of the studies were found to be at high risk of bias, with marked deficiencies in study design and outcome assessment.

A recent systematic review showed improved fascial closure rates with negative pressure wound therapy (NPWT) Yet, a large national study using NPWT to perform a DPC has been shown to actually decrease the rate of closure. Access to NPWT has increased over the years and innovative wound management techniques including incisional application of negative pressure therapy have allowed clinicians to apply this method to dirty wounds following the principles of delayed primary closure. There are currently no studies available to help determine the safety and efficacy of advanced NPWT techniques to optimize surgical wound management from the open abdomen to skin closure. Within our Division, we have decided to make a practice change and develop a standard closure plan for open abdomens using the negative pressure devices available within our institution.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* undergone midline laparotomy and managed with an open abdomen for at least one day
* contaminated or dirty wound classification

Exclusion Criteria:

* Less than 18 years of age
* Prisoners
* Pregnant females
* Non-surgical patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
30 day wound complication rate | 30 days
  Wound infection, dehiscence, evisceration
30 day readmission | 30 days
  Patient discharged and readmitted to primary care
Days of Abthera, VERAFLO, and Prevena use | through wound closure, an average of 30 days
  Use of negative pressure wound therapy
Closure of Fascia | 7 days
  Measure of days to closure of fascia
Closure of Skin | 7 days
  Measure of days to closure of skin
Cost of care | days to wound closure an average of 30 days
  Total cost for wound care

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States